CLINICAL TRIAL: NCT03883711
Title: Acute Myocardial Infarction From Clinical Presentation to Strategy Treatment
Brief Title: Acute Myocardial Infarction: Prognostic and Therapeutic Evaluation
Acronym: AMIPE
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Carmine Pizzi, Principal investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: 600/2018/Oss/AOUBo
Record Dates: First submitted 2019-03-15; First posted 2019-03-21 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Coronary Syndrome; Myocardium; Injury
Keywords: Acute coronary syndrome; Myocardial injury; ACS; MINOCA
MeSH Terms: conditions — Acute Coronary Syndrome; Wounds and Injuries; MINOCA | interventions — Database Management Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute coronary syndrome or myocardial injury: Incident consecutive patients presenting with acute coronary syndrome or myocardial injury
  Interventions: Other: Database

INTERVENTIONS:
Other: Database — Create a database containing clinical characteristic, clinical presentation, flow indexes and treatment of consecutive incident patients with ACS or myocardial injury.

SUMMARY:
AMIPE is both a retrospective and prospective study which was designed in order to collect data of patients with acute coronary syndromes and myocardial injury and to improve the knowledge about these conditions.

DETAILED DESCRIPTION:
AMIPE is an observational, multicenter and both retrospective and prospective study enrolling a cohort of consecutive incident patients admitted to participating hospitals with a diagnosis of acute coronary syndrome or myocardial injury from 01/01/2016 to 31/12/2023.

The aim of this study is to create a database including a comprehensive characterization of these patients in order to obtain new scientific evidence about these conditions. Informations about the patients will be gathered from in-hospital medical records. A written informed consent is needed for every prospective patients enrolled in the study,

In particular, the main objectives of the study are:

* document the characteristics of all patients presenting with acute coronary syndrome and myocardial injury;
* document the long term outcome rates;
* document the therapeutic regimens and investigation conformity of treatment with already established guidelines.

Every diagnostic or therapeutic intervention will be in accordance with established guidelines and good clinical practice.

Statistics will be conducted utilizing univariate and multivariate analysis for outcomes. In particular for what concerns univariate analysis, ordinal variables will be analysed with t-test and Mann-Whitney Test, whereas categorical responses with Fischer Exact Test and with Pearson Chi-square test.

Multivariate analysis will be conducted with logistic regression for dichotomous variables, with mixed generalized linear model for ordinal or nominal variables and with ANOVA or MANOVA for continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged > 18 years old
* Acute coronary syndrome or myocardial injury
* Written informed consent

Exclusion Criteria:

* under age or not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with a diagnosis of acute coronary syndrome or myocardial injury
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 1 year
  Death rate
All cause mortality | 3 years
  Death rate
All cause mortality | 5 years
  Death rate
Major Adverse Cardiac Events (MACEs) | 1 year
  MACEs rate
Major Adverse Cardiac Events (MACEs) | 3 years
  MACEs rate
Major Adverse Cardiac Events (MACEs) | 5 years
  MACEs rate

SECONDARY OUTCOMES:
Cardiovascular risk factors prevalence | 1 year
  Differences in percentage of patients with STEMI or NSTEMI, or type 1 or type 2 myocardial infarction with any risk factors
Cardiovascular risk factors prevalence | 3 year
  Differences in percentage of patients with STEMI or NSTEMI, or type 1 or type 2 myocardial infarction with any risk factors
Cardiovascular risk factors prevalence | 5 year
  Differences in percentage of patients with STEMI or NSTEMI, or type 1 or type 2 myocardial infarction with any risk factors
Differences in clinical presentation | 3 year
  Prevalence of patients presenting with ST elevation, angina, dyspnea, atypical chest pain, cardiogenic shock, arrhytmias)
Differences in clinical presentation | 1 year
  Prevalence of patients presenting with ST elevation, angina, dyspnea, atypical chest pain, cardiogenic shock, arrhytmias)
Differences in clinical presentation | 5 year
  Prevalence of patients presenting with ST elevation, angina, dyspnea, atypical chest pain, cardiogenic shock, arrhytmias)
Difference diagnosis between myocardial infarction subtypes and between myocardial infarction and myocardial injury | 5 year
  Differences in clinical presentation (ST elevation, angina, dyspnea, atypical chest pain, cardiogenic shock, arrhytmias)
Differences in flow characteristics | 1 year
  TIMI, TIMI frame count
Differences in flow characteristics | 3 year
  TIMI, TIMI frame count
Differences in flow characteristics | 5 year
  TIMI, TIMI frame count
Differences and impact of periprocedural ischemic complications | 5 year
  Type 4a myocardial infarction, periprocedural myocardial injury

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Pizzi, Dr, Principal Investigator — University of Bologna, Cardiology Department
Locations (3):
- Italy (3):
  - Policlinico Sant'Orsola-Malpighi, Cardiology Department, Bologna, Bologna
  - Ospedale Maggiore Carlo Alberto Pizzardi, Bologna, BO
  - Ospedale Morgagni - Pierantoni, Forlì, FC

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bonaca MP, Wiviott SD, Braunwald E, Murphy SA, Ruff CT, Antman EM, Morrow DA. American College of Cardiology/American Heart Association/European Society of Cardiology/World Heart Federation universal definition of myocardial infarction classification system and the risk of cardiovascular death: observations from the TRITON-TIMI 38 trial (Trial to Assess Improvement in Therapeutic Outcomes by Optimizing Platelet Inhibition With Prasugrel-Thrombolysis in Myocardial Infarction 38). Circulation. 2012 Jan 31;125(4):577-83. doi: 10.1161/CIRCULATIONAHA.111.041160. Epub 2011 Dec 23. PMID 22199016
- [Background] Sandoval Y, Smith SW, Sexter A, Thordsen SE, Bruen CA, Carlson MD, Dodd KW, Driver BE, Hu Y, Jacoby K, Johnson BK, Love SA, Moore JC, Schulz K, Scott NL, Apple FS. Type 1 and 2 Myocardial Infarction and Myocardial Injury: Clinical Transition to High-Sensitivity Cardiac Troponin I. Am J Med. 2017 Dec;130(12):1431-1439.e4. doi: 10.1016/j.amjmed.2017.05.049. Epub 2017 Jul 21. PMID 28739197
- [Background] Baron T, Hambraeus K, Sundstrom J, Erlinge D, Jernberg T, Lindahl B; TOTAL-AMI study group. Type 2 myocardial infarction in clinical practice. Heart. 2015 Jan;101(2):101-6. doi: 10.1136/heartjnl-2014-306093. Epub 2014 Oct 20. PMID 25331532
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Circulation. 2018 Nov 13;138(20):e618-e651. doi: 10.1161/CIR.0000000000000617. No abstract available. PMID 30571511
- [Derived] Canton L, Fedele D, Bergamaschi L, Foa A, Di Iuorio O, Tattilo FP, Rinaldi A, Angeli F, Armillotta M, Sansonetti A, Stefanizzi A, Amicone S, Impellizzeri A, Suma N, Bodega F, Cavallo D, Bertolini D, Ryabenko K, Casuso M, Belmonte M, Gallinoro E, Casella G, Galie N, Paolisso P, Pizzi C. Sex- and age-related differences in outcomes of patients with acute myocardial infarction: MINOCA vs. MIOCA. Eur Heart J Acute Cardiovasc Care. 2023 Sep 25;12(9):604-614. doi: 10.1093/ehjacc/zuad059. PMID 37261384
- [Derived] Paolisso P, Foa A, Bergamaschi L, Angeli F, Fabrizio M, Donati F, Toniolo S, Chiti C, Rinaldi A, Stefanizzi A, Armillotta M, Sansonetti A, Magnani I, Iannopollo G, Rucci P, Casella G, Galie N, Pizzi C. Impact of admission hyperglycemia on short and long-term prognosis in acute myocardial infarction: MINOCA versus MIOCA. Cardiovasc Diabetol. 2021 Sep 24;20(1):192. doi: 10.1186/s12933-021-01384-6. PMID 34560876